CLINICAL TRIAL: NCT05246423
Title: Paroxysmal Atrial Fibrillation Prognosis Based on Cardiopulmonary Exercise Test Data and Novel Echocardiographic and Plasma Biochemical Indices (the PLACEBO Trial)
Brief Title: Ergospirometry in Paroxysmal Atrial Fibrillation Prognosis
Acronym: PLACEBO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: General Hospital Of Thessaloniki Ippokratio (Other)
Responsible Party: Principal Investigator, Christodoulos Papadopoulos, Assistant Professor of Cardiology, Aristotle University Of Thessaloniki
Other Study IDs: 29551/30.6.2020
Record Dates: First submitted 2022-02-03; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation; Atrial Arrhythmia
Keywords: atrial fibrillation; cardiopulmonary exercise testing; exercise capacity; echocardiography; holter monitoring; peak oxygen uptake
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 40 ml plasma specimen (-80 grades Celcius)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: Patients with paroxysmal atrial fibrillation, recruited at least two weeks after the last paroxysm
  Interventions: Diagnostic Test: Observation group

INTERVENTIONS:
Diagnostic Test: Observation group — Patients with paroxysmal atrial fibrillation undergo cardiopulmonary exercise testing, echocardiography, 24-hour ambulatory electrocardiographic monitoring and plasma biomarkers' measurement

SUMMARY:
An observational, prospective, cohort study aiming to assess the potential predictive role of cardiopulmonary exercise testing in the prognosis of paroxysmal atrial fibrillation, in combination with echocardiographic indices and plasma biomarker values.

DETAILED DESCRIPTION:
The "ParoxysmaL Atrial fibrillation prognosis based on Cardiopulmonary Exercise test data and novel echocardiographic and plasma BiOchemical indices" (PLACEBO) trial comprises an observational, prospective, single-center cohort study including patients with paroxysmal atrial fibrillation. All patients undergo clinical examination, detailed echocardiographic study, cardiopulmonary exercise testing (CPET) and 24-hour ambulatory echocardiographic monitoring (24-hour Holter monitoring), as well as measurement of a series of plasma biochemical indices. The study will examine the potential prognostic role of CPET variables (such as peak VO2) in the future recurrences of paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with paroxysmal atrial fibrillation (in sinus rhythm during baseline evaluation)
2. Age > 18 years
3. Capability of providing written consent
4. Patients able to undergo cardiopulmonary exercise testing
5. Patients able to comply with the follow-up schedule of the study

Exclusion Criteria:

1. Patients with structural cardiomyopathy
2. Patients with congenital heart disease
3. Patients with permanent atrial fibrillation
4. Patients who have undergone atrial fibrillation ablation
5. Patients with implanted cardiac devices for primary or secondary prevention
6. Patients with recent (within the last month) acute coronary syndrome
7. Patients with heart failure with reduced ejection fraction (HFrEF) or end-stage renal disease
8. Patients with autoimmune diseases or active malignancies
9. Patients with uncontrolled thyroid disease
10. Patients unable to undergo cardiopulmonary exercise testing due to disability or motility issues
11. Patients who present with contraindications for cardiopulmonary exercise testing
12. Patients unable to provide written consent
13. Patients with poor echocardiographic images
14. Patients unable to undergo spirometry
15. Patients unable to comply with the follow-up schedule of the study
16. Patients with uncontrolled hypertension
17. Patients who have undergone recent (within the last 2 months) surgery
18. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal atrial fibrillation, at least 2 weeks after the last atrial fibrillation episode, are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of new atrial fibrillation paroxysms | 2 months
  The primary outcome of the study is the total number of atrial fibrillation paroxysms within one year of baseline visit.
Number of new atrial fibrillation paroxysms | 6 months
  The primary outcome of the study is the total number of atrial fibrillation paroxysms within one year of baseline visit.
Number of new atrial fibrillation paroxysms | 12 months
  The primary outcome of the study is the total number of atrial fibrillation paroxysms within one year of baseline visit.

SECONDARY OUTCOMES:
Atrial fibrillation - related hospitalizations | 2 months - 6 months - 12 months
  The total number of atrial fibrillation - related hospitalizations
Type of cardioversions | 2 months - 6 months - 12 months
  In case of new atrial fibrillation paroxysms, the total number and type of cardioversions (electrical, pharmaceutical, spontaneous)
Total burden of premature atrial contractions | Baseline and 12 months
  Total number of premature atrial contractions recorded during the 24-hour ambulatory electrocardiographic monitoring
Total burden of premature ventricular contractions | Baseline and 12 months
  Total number of premature atrial contractions recorded during the 24-hour ambulatory electrocardiographic monitoring
Atrial fibrillation episodes during 24-hour ambulatory electrocardiographic monitoring | Baseline and 12 months
  Total atrial fibrillation episodes recorded 24-hour ambulatory electrocardiographic monitoring
Microvolt T-wave Alternans (TWA) | Baseline and 12 months
  Specialist software quantifies microvolt TWA voltage in patients' 24-hour ambulatory electrocardiographic monitor recordings
Heart rate turbulence (HRT) | Baseline and 12 months
  Heart rate turbulence (HRT) is the baroreflex-mediated short-term oscillation of cardiac cycle lengths after spontaneous ventricular premature complexes. Specialist software detects abnormal HRT in patients' 24-hour ambulatory electrocardiographic monitor recordings
Deceleration capacity (DC) | Baseline and 12 months
  (Heart rate) deceleration capacity is a measurement of autonomic nerve regulation in heart failure. Specialist software quantifies deceleration capacity, which is measured in milliseconds (ms).
Peak oxygen uptake (peak VO2) | Baseline
  Peak oxygen uptake values, measured in ml/kg/min during cardiopulmonary exercise testing
Minute ventilation/carbon dioxide production slope (VE/VCO2 slope) | Baseline
  Minute ventilation/carbon dioxide production slope (VE/VCO2 slope) measured during cardiopulmonary exercise testing
Left atrial strain | Baseline and 12 months
  Left atrial strain measured during echocardiographic study
Left ventricular global longitudinal strain (GLS) | Baseline and 12 months
  Left ventricular global longitudinal strain (GLS) measured during echocardiographic study
Plasma biomarkers | Baseline and 12 months
  Values of plasma biomarkers (GDF-15, IL-6, hs-cTnI)
Time to first recurrence | 12 months
  Time from baseline to first recurrence of atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Aristi C. Boulmpou, MSc, Principal Investigator — Aristotle University of Thessaloniki, Greece; Christodoulos E. Papadopoulos, PhD, Principal Investigator — Aristotle University of Thessaloniki, Greece
Locations (1):
- Ippokratio General Hospital, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided